CLINICAL TRIAL: NCT02155426
Title: A Multicenter, Prospective, Observational Trial on the Prognostic and Dynamic Change of CTC Enumeration in Advanced NSCLC With 1st or 2nd Line Line Chemotherapy and Targeted Therapy
Brief Title: Prognostic and Dynamic Change of CTC Enumeration in Advanced NSCLC With Chemotherapy and Targeted Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cyttel Biosciences Inc. (Industry)
Responsible Party: Principal Investigator, Li Zhang, Head of GCP, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Other Study IDs: NSCLCCTC-SUMS01
Record Dates: First submitted 2014-05-13; First posted 2014-06-04 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Subjects' blood sample will be retained to evaluate the dynamic CTC count during the treatment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment: Treatment: Chemotherapy or targeted therapy

SUMMARY:
TITLE : A Multicenter, Prospective, Observational Trial on the Prognostic and Dynamic Change of CTC Enumeration in Advanced NSCLC with 1st or 2nd line chemotherapy and targeted therapy

BACKGROUND : Circulating tumor cells (CTC) identification is a new field of research in oncology, and some studies have been conducted with success on breast and prostate cancer. Nearly 80% of lung cancers are diagnosed in an advanced stage (IIIB, and IV). CTC identification and monitoring these cells after treatment could help the clinicians to detect relapse or be a prognostic factor.

PRIMARY OBJECTIVE : To study the relationship between CTC count and clinical outcome of treatment (Overall response rate and Progression-free survival).

SECONDARY OBJECTIVES :To study the relationship between CTC and overall survival.

STUDY DESIGN : This is a prospective, observational study.

Duration of the inclusions: 12months.

SAMPLE SIZE : 1200 patients

DETAILED DESCRIPTION:
This is a prospective observational non-intervention study evaluating the dynamic CTC count during the chemotherapy and targeted-therapy. Patients provide written informed consent and pass the screening. Peripheral blood will be drawn before and after the treatment. Relationship between CTC count and clinical outcome will be analysed. The time points of blood drawing are set as following: for patients receiving chemotherapy, once prior to 1st cycle of chemotherapy, once 3 days prior to 2nd cycle of chemotherapy, posterior to 3th cycle (or less than 4th cycle) of chemotherapy and once when progressive disease (PD); for patients receiving targeted-therapy, once prior to treatment, once 1 month after treatment, and once when PD. The clinical outcome of treatment will be ultimately obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented, locally advanced or recurrent (stage IIIb and not amenable or combined modality treatment) or metastatic (stage IV) non-small cell lung cancer.
* ECOG functional status≤2
* Chemotherapy:According to routine 1st line doublet chemotherapy in clinical practice, Cisplatin or carboplatin combined with gemcitabine or paclitaxel or docetaxol or Vinorelbine were recommended. According to routine 2nd line chemotherapy in clinical practice,pemetrexed or docetaxol
* Targeted therapy：According to clinical criteria, patients with EGFR-TKI sensitive mutant accept first line TKI therapy.
* Patients must have measurable disease according to the RECIST (version 1.1) criteria
* Patients with a life expectancy greater than 12 weeks
* Written (signed) informed Consent to participate in the study

Exclusion Criteria:

* Patients with history of any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids.
* Unwilling to write informed consent to participate in the study
* Patients who is unwilling to accept the follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically documented, locally advanced or recurrent (stage IIIb and not amenable or combined modality treatment) or metastatic (stage IV) non-small cell lung cancer, who will receive routine first or second line chemotherapy, or EGFR-TKI for those with EGFR sensitive mutant type.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Baseline CTC count | Two year

SECONDARY OUTCOMES:
CTC count change | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China